CLINICAL TRIAL: NCT01703195
Title: Magnetic Resonance Imaging of Gynecologic Malignancies Involving the Vagina
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2011-0656; NCI-2012-02054 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2012-10-05; First posted 2012-10-10 (Estimated); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Vaginal Cancer
Keywords: Vaginal Cancer; Malignancies involving the vagina; Middle third and the distal third of the vagina; Pre and post radiation therapy; Diffusion weighted magnetic resonance imaging; DWMR; Magnetic resonance imaging; MRI; Tumor involvement; Response to radiation therapy; XRT
MeSH Terms: conditions — Vaginal Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Diffusion Weighted Magnetic Resonance Imaging (DWMR) (Other): Patients receive Magnetic Resonance Imaging (MRI) and Diffusion Weighted Magnetic Resonance Imaging (DWMR) imaging pre-treatment and 4-6 weeks post-treatment.
  Interventions: Procedure: Magnetic Resonance Imaging (MRI); Procedure: Diffusion Weighted Magnetic Resonance Imaging (DWMR)

INTERVENTIONS:
Procedure: Magnetic Resonance Imaging (MRI) — Magnetic Resonance Imaging (MRI) obtained pre-treatment and 4-6 weeks post-treatment.
  Other Names: MRI
Procedure: Diffusion Weighted Magnetic Resonance Imaging (DWMR) — Diffusion Weighted Magnetic Resonance Imaging (DWMR) obtained pre-treatment and 4-6 weeks post-treatment.
  Other Names: DWMR

SUMMARY:
The goal of this clinical research study is to learn if a type of MRI scan called diffusion weighted imaging (DWI) is accurate in checking the status of tumors. Researchers also want to learn if DWI can predict how tumors will respond to radiation therapy.

DETAILED DESCRIPTION:
If you agree to take part in this study, information will be collected from your medical record including your age, sex, and status of the disease.

For the MRI scans, you will receive a routine contrast drug by vein. Contrast drugs are used by doctors in order to see MRI images more clearly.

A modified MRI scan will performed right after your scheduled standard-of-care MRI scan. This modified MRI scan is the investigational scan. To complete the modified MRI scan, you will need to stay in the MRI scanner for about 8 extra minutes. It should take about 47 minutes total to complete both scans.

The way that researchers program the MRI machine and the order in which the images are taken is what is being modified for the investigational scan. These changes may help researchers capture better images.

Length of Study:

Your participation on this study will be over after the modified MRI scan is complete.

This is an investigational study. The standard-of-care MRI scan method is FDA approved and commercially available for the diagnosis of several diseases. The modified MRI scan method is being used in research only.

Up to 25 participants will be enrolled in this study. All will take part at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. All patients who have gynecologic malignancies involving the middle third and the distal third of the vagina who will be receiving radiation therapy
2. Patients who have gynecologic malignancies involving the upper, middle and/or lower third of the vagina or are undergoing pelvic exenteration.

Exclusion Criteria:

1. Pregnant patients
2. Any implantable medical device that is not MRI compatible (e.g. pacemakers, defibrillators, pain pumps or insulin pumps)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2019-09-19 (Actual); Study Completion 2019-09-19 (Actual)

PRIMARY OUTCOMES:
Accuracy of Tumor Involvement Detection | 1 day
  Location of tumor involvement determined based on pre-treatment imaging findings, where inferior margin of tumor marked on the MRI. Tumor involved areas will then be evaluated by EUA, where fiducial markers will be placed and MRI images will be fused with the CT images to find if there is any discrepancy between the EUA and the DWI images. The primary endpoint is the accuracy of tumor involvement detection (binary endpoint), where tumor invasion is defined as similar to that seen by EUA, in the anterior/posterior or the lateral walls of the vagina. Similarity will be defined as the tumor margin seen on MRI being similar to what is seen on the EUA where the markers correspond to the margins defined on the MRI. This will be defined as 5mm or less.

SECONDARY OUTCOMES:
Ability of Diffusion Weighted Magnetic Resonance Imaging (DWMR) to Assess Response to Radiation Therapy | 4 weeks after radiation therapy treatment
  Secondary endpoints include quantitative measurements of discrepancies (or: quantitative measurement of the discrepancy) between DWMR and exam under anesthesia (EUA), agreement and difference between DWMR and other MR sequences (T2, DGE), and the ability of DWMR to assess response to therapy. Summary statistics of results for each modality tabulated. Accuracy, sensitivity, specificity, PPV, and NPV estimated along with corresponding 95% CIs. Quantitative discrepancy measurements summarized using mean, SD, and range. Difference and agreement between DWMR and other MR sequences assessed using the McNemar test and Kappa statistics, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Priya Bhosale, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org